CLINICAL TRIAL: NCT00665548
Title: Weight-Bearing MRI for Analysis of Knee OA
Brief Title: Weight-Bearing Magnetic Resonance Imaging (MRI) for Analysis of Knee Osteoarthritis (OA)
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sharmila Majumdar, PhD, UCalifroniaSF
Other Study IDs: Pfizer West
Record Dates: First submitted 2008-04-22; First posted 2008-04-24 (Estimated); Last update posted 2009-04-17 (Estimated); Status verified 2008-03

CONDITIONS: Osteoarthritis
Keywords: Knee Osteoarthritis; magnetic resonance imaging; x rays
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — X-Rays; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (2):
- Normal Subjects: Female subjects scoring Kellgren & Lawrence grade 0.
  Interventions: Radiation: X-ray; magnetic resonance imaging
- OA Subjects: Female subjects with Kellgren & Lawrence score of 2 or 3.
  Interventions: Radiation: X-ray; magnetic resonance imaging

INTERVENTIONS:
Radiation: X-ray; magnetic resonance imaging — Knee x-rays: acquired in both a standard or weight-bearing position and in non-weight-bearing position to measure joint space width and look at signs of osteoarthritis.
  3 Tesla MRI: magnetic resonance imaging of the study knee during weight-bearing conditions and traditional non-loaded condition all acquired with the same sequences.

SUMMARY:
The purpose of the study is to use different x-ray and magnetic resonance (MR) imaging techniques to take pictures of the knee. There are two specific purposes to the study:

1. whether the different x-ray and MRI techniques will give the same or different information about the knee joint and
2. which part of the knee joint will show the biggest change using the different x-ray and MRI techniques. The study is not designed to test a hypothesis.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 40 years and older
* Subjects who are willing and able to comply with x-ray and MRI procedures
* Evidence of a personally signed and dated consent document

Additional inclusion for normal controls:

* Infrequent knee pain, aching, or stiffness during the past year or infrequent use of medication for treatment of knee pain during the past year
* No evidence of OA on either knee (i.e. K-L grade = 0 diagnosed by knee radiography)

Additional inclusion for OA patients:

* Pain, aching, or stiffness on most days of a month during the past year; or use of medication for treatment of knee pain on most days of a month during the past year
* Kellgren-Lawrence Grade 2 or 3 of the study knee obtained on a Standard knee radiograph (with either the same or less severe OA, or no OA in the contralateral knee)

Exclusion Criteria:

* Subject is unable to undergo MRI because of contraindication
* Women at risk of pregnancy
* Weight greater than 250 lbs
* History of surgery in the study knee
* History of other diseases involving the study knee joint including inflammatory joint diseases, crystalline disease, and infection of the study knee

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female, 40 years and older, community sample
Sampling Method: Non-Probability Sample
Enrollment: 33 (Estimated)
Dates: Start 2008-03; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Determine which joint components demonstrate the greatest changes between weight-bearing and non weight-bearing protocols. | at time of scan

SECONDARY OUTCOMES:
Determine if additional information gained from weight-bearing images can explain the difference in joint space width (JSW) between weight-bearing x-ray and traditional non-weight bearing MRI. | at time of scan

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Majumdar, PhD, Principal Investigator — University of California, San Francisco; Thomas Link, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California - San Francisco, San Francisco, California, United States